CLINICAL TRIAL: NCT00583765
Title: Evaluation of a Simplified Protocol for Regional Citrate Anticoagulation in Continuous Venovenous Hemodiafiltration
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Gambro Renal Products, Inc. (Industry)
Responsible Party: R.T.Noel Gibney, Division of Critical Care Medicine, University of Alberta
Other Study IDs: 5793
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Kidney Failure, Acute
Keywords: Kidney Failure, Acute; Hemodialysis; Hemofiltration; Anticoagulation; Citrate
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Critically ill patients with acute renal failure requiring continuous renal replacement therapy
  Interventions: Drug: Regional citrate anticoagulation

INTERVENTIONS:
Drug: Regional citrate anticoagulation — Continuous venovenous hemodiafiltration with regional anticoagulation using dilute trisodium citrate. This requires the use of a continuous renal replacement therapy (CRRT) machine in venovenous hemodiafiltration mode. Anticoagulation and buffer are provided by the use of a dilute solution of trisodium citrate in the replacement fluid which is infused in a predilution mode. Standard bicarbonate containing dialysate is used.
  Other Names: Prismocitrate - the study fluid; Prismocal - the commercially available dialysate

SUMMARY:
Dialysis requires thinning of the blood to prevent clotting in the dialysis machine. Thinning of the blood is necessary but some forms of blood thinners may cause bleeding. Therefore, researchers are seeking ways to minimize bleeding risks and ensure effective dialysis.

One medication used to thin the blood in the dialysis machine is citrate. Citrate has the advantage of having its blood-thinning properties quickly reversed by calcium in the patient's blood. As a consequence, only the blood in the machine is thinned, greatly reducing the risk of bleeding when dialysis is carried out using other blood thinners. Until now, most patients who received citrate for dialysis were administered the citrate in a separate infusion through an IV pump into the dialysis machine. This method requires complex monitoring and calculations. This study is about Prismocitrate which is a dialysis fluid very similar to the regular dialysis fluid that is used in this intensive care unit, except that this fluid already contains exactly the correct amount of citrate. Thus, this method does not require a separate pump for citrate and calculations to pump the citrate into the blood as it goes through the kidney machine. Having the citrate already contained in the dialysis fluid simplifies the procedure and reduces the possibility of calculation errors.

This study seeks to determine if this simplified means of providing blood thinning in the kidney machine also results in the correct balance of blood salts.

DETAILED DESCRIPTION:
Acute renal failure is common among the critically ill [1-3] , and is an independent contributor to morbidity and mortality [4,5]. Continuous renal replacement therapy (CRRT) is commonly used for renal replacement in this group. This requires an extracorporeal circuit, the maintenance of which requires anticoagulation. Heparin has been the most common anticoagulant used with CRRT. However, heparin exposure for CRRT is major risk after surgery or trauma. Citrate has been used as a regional anticoagulant for plasmapheresis and chronic dialysis for many years [12,13], and is increasingly being used for CRRT. Regional anticoagulation refers to the provision of anticoagulation within the extracorporeal circuit without any alteration in coagulation in the patient's systemic circulation. Calcium is a co-factor in coagulation. Citrate reduces levels of ionized calcium in blood of the extracorporeal circuit to levels where coagulation cannot occur. Once the blood is returned to the patient's systemic circulation, the calcium levels are restored and coagulation can occur again. Renal replacement solutions for CRRT using citrate anticoagulation, should be calcium-free. [14-19] Despite a reduced risk of bleeding, widespread adoption of citrate regional anticoagulation has been limited by a lack of commercially available calcium-free solutions and the complexity of many protocols. Part of this complexity is the requirement for a separate citrate infusion into the extracorporeal circuit to achieve regional anticoagulation. This simplified protocol provides citrate in the replacement fluid infused prefilter as both anticoagulant and as buffer.

To predict appropriate replacement rates, Hospal Gambro scientific laboratories have developed a calculation model to predict the physiological interactions between the components of the administered replacement- and hemodialysis fluids and the patient's complex metabolic system. These interactions are influenced, in large part, by systemic parameters such as blood-flow and ultrafiltration rates, and patient parameters, such as acid base-status and liver function. This calculation model needs clinical validation in respect to its ability to predict the outcome and narrow the margin of metabolic disturbances caused by the administration of citrate anticoagulation. A previous study of a similar replacement fluid using citrate 8 mmol/L and citric acid 4 mmol/L resulted in mild metabolic acidosis of minimal clinical significance in some subjects and so this study will evaluate a modified version of fluid containing citrate 10 mmol/L and citric acid 2 mmol/L which has been calculated to provide optimal metabolic balance.

Subjects:

Twenty patients in the General Systems ICU at the University of Alberta Hospital treated with CVVHDF using a Prisma-CFM machine will be studied.

Inclusion criteria:

1. Male or female between 17 and 80 years of age.
2. Intensive care unit patient.
3. Renal failure requiring CVVHDF.
4. Likely to survive for at least 72 hours.

Exclusion criteria

1. Age > 80 years
2. Need for systemic anticoagulation, fibrinolytic therapy or activated protein C
3. Acute or chronic hepatic failure

Patients are treated by regular CVVHDF setting in pre-dilution mode. The replacement flow-rate for the citrate replacement fluid depends on the blood pump speed [fixed ratio, see 9.3 and table below]. Mean dialysate flow is between 100 ml/hr and 2500ml/hour in accordance to the desired base-equivalent intake. Access pressure is kept between -100 and 150mmHg. Access and return pressure are monitored. Specially formulated replacement- and dialysate fluids are used.

Citrate anticoagulation Published literature data show that a mean citrate-dosage of 3.5 to 4mmol/l of undiluted blood is necessary to decrease the level of ionized serum calcium below 0.4mmol/l which provides sufficient anticoagulation to maintain an extracorporeal circuit. A minimum citrate concentration of 3.5 mmol/l blood will be used in this protocol. The infused citrate replacement fluid contains trisodium citrate and citric acid in a mixture (10mmol/l tri-sodium citrate plus 2 mmol/l citric acid). Preliminary results proved that the anticoagulation potency of this mixture is similar to a plain 12 mmol/l tri-sodium citrate solution. Therefore a fixed ratio of citrate replacement fluid will be infused in pre-pump predilution mode per 1 liter of effective blood flow.

Calcium replacement:

The loss of calcium- and magnesium-citrate in the ultra-filtrate via the hemofilter needs to be compensated to avoid systemic hypocalcemia and hypomagnesemia. Calcium replacement solution is prepared by removing 300 mls from a 1000 mls bag of 0.9% saline and subsequently adding 200 mls of 10% calcium gluconate to this bag. This calcium gluconate solution is infused via a central line at an initial infusion rate of 60 ml/hr. Ionized calcium levels are monitored every 6-8 hours and corrected by changing of flow rate of the infusion.

Potassium replacement:

Potassium is added into the replacement and dialysate fluid based on clinical requirement.

Sodium-bicarbonate adjustment:

The sodium bicarbonate level is influenced by the flow-rate of the replacement fluid (citrate intake) and the dialysate flow (bicarbonate intake). It is monitored every 6 hours and is corrected during treatment by altering the dialysate flow. Reducing the flow rate lowers bicarbonate intake in case of metabolic alkalosis, raising flow increases the bicarbonate intake in case of metabolic acidosis. If these adjustments are not successful, further corrections can be done by adding bicarbonate into the next dialysate fluid bag, when it is changed:

Consent procedure Subjects will be identified, recruited and informed consent obtained by the principal investigator, co-investigator or research co-ordinators.

Study benefits The study renal replacement solution includes all elements required for safe use. It does not require custom preparation by hospital personnel. This will minimize risk of error and increase patient safety. It is hoped this study will eventually enable the general use of a simple safe technique for citrate regional anticoagulation during continuous renal replacement therapy.

Adverse effects CVVHDF using citrate regional anticoagulation using any protocol may be associated with hypocalcemia, metabolic alkalosis or acidosis, hypernatremia or hyponatremia. In anticipation of this, all protocols including this one use extensive metabolic monitoring and algorithmic responses to abnormalities. This simplified protocol minimizes the potential for complication.

Adverse effects would be notified to patient or family, investigator, and HREB committee.

Privacy Patient data will be anonymized to prevent identification. Gambro Canada (study sponsor) will have access to anonymized case report forms and aggregate report.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 17 and 80 years of age.
* Intensive care unit patient.
* Acute renal failure requiring continuous venovenous hemodiafiltration.
* Likely to survive for at least 72 hours

Exclusion Criteria:

* Age > 80 years
* Need for systemic anticoagulation, fibrinolytic therapy or activated protein C
* Acute or chronic hepatic failure

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Male or female between 17 and 80 years of age.
  2. Critically ill intensive care unit patient.
  3. Renal failure requiring continuous venovenous hemodiafiltration.
  4. Likely to survive for at least 72 hours
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
metabolic stability | 24, 48 and 72 hours

SECONDARY OUTCOMES:
Hemofilter survival | 24, 48 and 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Noel Gibney, MB BCh BAO, Principal Investigator — University of Alberta
Locations (1):
- General Systems Intensive Care Unit, University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Uchino S, Kellum JA, Bellomo R, Doig GS, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Ronco C; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Acute renal failure in critically ill patients: a multinational, multicenter study. JAMA. 2005 Aug 17;294(7):813-8. doi: 10.1001/jama.294.7.813. PMID 16106006
- [Background] Tolwani AJ, Campbell RC, Schenk MB, Allon M, Warnock DG. Simplified citrate anticoagulation for continuous renal replacement therapy. Kidney Int. 2001 Jul;60(1):370-4. doi: 10.1046/j.1523-1755.2001.00809.x. PMID 11422774
- [Background] Uchino S, Bellomo R, Kellum JA, Morimatsu H, Morgera S, Schetz MR, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Oudemans-Van Straaten HM, Ronco C; Beginning and Ending Supportive Therapy for the Kidney (B.E.S.T. Kidney) Investigators Writing Committee. Patient and kidney survival by dialysis modality in critically ill patients with acute kidney injury. Int J Artif Organs. 2007 Apr;30(4):281-92. doi: 10.1177/039139880703000402. PMID 17520564
- [Background] Tolwani AJ, Prendergast MB, Speer RR, Stofan BS, Wille KM. A practical citrate anticoagulation continuous venovenous hemodiafiltration protocol for metabolic control and high solute clearance. Clin J Am Soc Nephrol. 2006 Jan;1(1):79-87. doi: 10.2215/CJN.00040505. Epub 2005 Nov 23. PMID 17699194
- [Background] Kutsogiannis DJ, Gibney RT, Stollery D, Gao J. Regional citrate versus systemic heparin anticoagulation for continuous renal replacement in critically ill patients. Kidney Int. 2005 Jun;67(6):2361-7. doi: 10.1111/j.1523-1755.2005.00342.x. PMID 15882280
- [Background] Kutsogiannis DJ, Mayers I, Chin WD, Gibney RT. Regional citrate anticoagulation in continuous venovenous hemodiafiltration. Am J Kidney Dis. 2000 May;35(5):802-11. doi: 10.1016/s0272-6386(00)70248-4. PMID 10793012
- [Background] Jacka MJ, Ivancinova X, Gibney RT. Continuous renal replacement therapy improves renal recovery from acute renal failure. Can J Anaesth. 2005 Mar;52(3):327-32. doi: 10.1007/BF03016071. PMID 15753507
- [Background] Gibney RT, Kimmel PL, Lazarus M. The Acute Dialysis Quality Initiative--part I: definitions and reporting of CRRT techniques. Adv Ren Replace Ther. 2002 Oct;9(4):252-4. doi: 10.1053/jarr.2002.35571. PMID 12382226
- [Background] Gibney RT, Stollery DE, Lefebvre RE, Sharun CJ, Chan P. Continuous arteriovenous hemodialysis: an alternative therapy for acute renal failure associated with critical illness. CMAJ. 1988 Nov 1;139(9):861-6. PMID 3179891
- [Background] Morath C, Miftari N, Dikow R, Hainer C, Zeier M, Morgera S, Weigand MA, Schwenger V. Sodium citrate anticoagulation during sustained low efficiency dialysis (SLED) in patients with acute renal failure and severely impaired liver function. Nephrol Dial Transplant. 2008 Jan;23(1):421-2. doi: 10.1093/ndt/gfm629. Epub 2007 Oct 3. No abstract available. PMID 17913732
- [Background] Fischer KG. Essentials of anticoagulation in hemodialysis. Hemodial Int. 2007 Apr;11(2):178-89. doi: 10.1111/j.1542-4758.2007.00166.x. PMID 17403168
- [Background] Amanzadeh J, Reilly RF Jr. Anticoagulation and continuous renal replacement therapy. Semin Dial. 2006 Jul-Aug;19(4):311-6. doi: 10.1111/j.1525-139X.2006.00178.x. PMID 16893409
- [Background] Mariano F, Tetta C, Ronco C, Triolo G. Is there a real alternative anticoagulant to heparin in continuous treatments? Expert Rev Med Devices. 2006 Jan;3(1):5-8. doi: 10.1586/17434440.3.1.5. No abstract available. PMID 16359246
- [Background] Gritters M, Grooteman MP, Schoorl M, Schoorl M, Bartels PC, Scheffer PG, Teerlink T, Schalkwijk CG, Spreeuwenberg M, Nube MJ. Citrate anticoagulation abolishes degranulation of polymorphonuclear cells and platelets and reduces oxidative stress during haemodialysis. Nephrol Dial Transplant. 2006 Jan;21(1):153-9. doi: 10.1093/ndt/gfi069. Epub 2005 Sep 6. PMID 16144857
- [Background] Gabutti L, Ferrari N, Mombelli G, Keller F, Marone C. The favorable effect of regional citrate anticoagulation on interleukin-1beta release is dissociated from both coagulation and complement activation. J Nephrol. 2004 Nov-Dec;17(6):819-25. PMID 15593057
- [Background] Morgera S, Scholle C, Voss G, Haase M, Vargas-Hein O, Krausch D, Melzer C, Rosseau S, Zuckermann-Becker H, Neumayer HH. Metabolic complications during regional citrate anticoagulation in continuous venovenous hemodialysis: single-center experience. Nephron Clin Pract. 2004;97(4):c131-6. doi: 10.1159/000079171. PMID 15331942
- [Background] Mariano F, Tetta C, Stella M, Biolino P, Miletto A, Triolo G. Regional citrate anticoagulation in critically ill patients treated with plasma filtration and adsorption. Blood Purif. 2004;22(3):313-9. doi: 10.1159/000078788. PMID 15256798
- [Background] Swartz R, Pasko D, O'Toole J, Starmann B. Improving the delivery of continuous renal replacement therapy using regional citrate anticoagulation. Clin Nephrol. 2004 Feb;61(2):134-43. doi: 10.5414/cnp61134. PMID 14989634
- [Background] Bunchman TE, Maxvold NJ, Brophy PD. Pediatric convective hemofiltration: Normocarb replacement fluid and citrate anticoagulation. Am J Kidney Dis. 2003 Dec;42(6):1248-52. doi: 10.1053/j.ajkd.2003.08.026. PMID 14655197
- [Background] Tobe SW, Aujla P, Walele AA, Oliver MJ, Naimark DM, Perkins NJ, Beardsall M. A novel regional citrate anticoagulation protocol for CRRT using only commercially available solutions. J Crit Care. 2003 Jun;18(2):121-9. doi: 10.1053/jcrc.2003.50006. PMID 12800123
- [Background] Gabutti L, Marone C, Colucci G, Duchini F, Schonholzer C. Citrate anticoagulation in continuous venovenous hemodiafiltration: a metabolic challenge. Intensive Care Med. 2002 Oct;28(10):1419-25. doi: 10.1007/s00134-002-1443-y. Epub 2002 Sep 6. PMID 12373466
- [Background] Bunchman TE, Maxvold NJ, Barnett J, Hutchings A, Benfield MR. Pediatric hemofiltration: Normocarb dialysate solution with citrate anticoagulation. Pediatr Nephrol. 2002 Mar;17(3):150-4. doi: 10.1007/s00467-001-0791-0. PMID 11956849
- [Background] Palsson R, Laliberte KA, Niles JL. Choice of replacement solution and anticoagulant in continuous venovenous hemofiltration. Clin Nephrol. 2006 Jan;65(1):34-42. doi: 10.5414/cnp65034. PMID 16429840
- [Background] Palsson R, Niles JL. Regional citrate anticoagulation in continuous venovenous hemofiltration in critically ill patients with a high risk of bleeding. Kidney Int. 1999 May;55(5):1991-7. doi: 10.1046/j.1523-1755.1999.00444.x. PMID 10231464
- [Background] Ward DM. The approach to anticoagulation in patients treated with extracorporeal therapy in the intensive care unit. Adv Ren Replace Ther. 1997 Apr;4(2):160-73. doi: 10.1016/s1073-4449(97)70043-8. PMID 9113232
- [Background] Ward DM, Mehta RL. Extracorporeal management of acute renal failure patients at high risk of bleeding. Kidney Int Suppl. 1993 Jun;41:S237-44. PMID 8320930